CLINICAL TRIAL: NCT00466154
Title: The Effect of Serum LDL Lowering on Aspirin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziv Hospital (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP 5-173 S
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Aspirin Resistance; Hypercholesterolemia
Keywords: Aspirin resistance; Platelet activation; Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Aspirin

SUMMARY:
Aspirin resistance is the persistent platelet activation, demonstrated by platelet function tests (1).

The hypothesis is that:LDL lowering by statin in patients with aspirin resistance can improve the effect of aspirin due to the potential decreasing of cholesterol content in the platelet membranes.

Patients and methods:Forty hypercholesterolemic patients with aspirin resistance after 5 days of treatment with aspirin and high LDL and triglycerides<300 mg/dL, will be enrolled.

Ten healthy volunteers will be the control group.

DETAILED DESCRIPTION:
The patients will be treated by aspirin loading dose of 500mg and then 100 mg/day for other 4 days. For patients that will be entrolled in the regular working hours, platelet aggregation test and cholesterol content in platelet membranes will be done at baseline.

Blood tests for lipids, liver (ALT,AST,GGT,Alkaline phosphatase and bilirubin) and renal function tests (blood urea nitrogen and creatinine), complete blood count, general urine test and serum homocysteine will be done on the second day.

On the fifth day optical platelet aggregation test, cholesterol content in platelet membranes, platelet function in the PFA-100 system and soluble p-selectin in the plasma will be done If the patient has aspirin resistance (platelet aggregation 20% with epinephrine or 70% with ADP), LDL will be lowered in the plasma of 20 patients by hypolipidemic drugs (statin alone or combined with ezetimibe). Other 20 patients will continue to be treated by aspirin alone.

One month later, blood tests for lipids, liver (ALT,AST,GGT,Alkaline phosphatase and bilirubin) and renal function tests (blood urea nitrogen and creatinine), complete blood count, general urine test and serum homocysteine will be done for the second time and platelet activity will be tested again for all patients.

Platelet separation:

For platelet studies, venous blood (30 ml) will be collected through siliconized syringes into acid citrate dextrose solution(1.4% citric acid, 2.5% sodium citrate, and 2% dextrose) at a ratio of 9:1 (v:v) for washed platelets (WP)preparation.WP will be prepared by centrifugation at 240g for 20 min. The platelet bellet will be washed twice in 5 mmol Hepes buffer, pH 7.4 (140 mmol NaCl, 2 mmol KCL, 1 mmol MgCl2, 5 mmol Hepes, 12 mmol NaHCO3 and 5.5 mmol of glucose). For the preparation of WP suspension, 15 uL of acetic acid (1mmol) will be added to 1 ml of platelet suspension throughout WP preparation in order to ensure acidic conditions which are required for platelet resuspension. This procedure will reduce the medium pH to 6.5 and it does not influence the aggregation response of the WP.

Platelet aggregation:

Collagen (Nycomed, germany) will be used as the aggregating agent at a concentration of 4 ug/ml (this concentration can cause up to 60% aggregation amplitude in WP). Platelet aggregation will be perfomed at 37ºC in aggregometer using hepes as a reference system. Results will be expressed as the extent of maximal aggregation (% of maximal amplitude) and also as the slope of the aggregation curve (cm/min).

Cholesterol content in platelet membranes:

Platelets will be washed three times with Hepes buffer, and then sonicated twice for 20 seconds at 80 watt. Platelet lipids will be extracted with hexane:isopropanolol (3:2, v:v). The cholesterol content will be measured in the dried hexane phase by the method of Chiamori et al (12). Platelet protein will be determined using the method of Lowry (13).

ELIGIBILITY:
Inclusion Criteria:

1. Hypercholesterolemic low-moderate risk patients without hypolipidemic drugs for at least one month.
2. Age ≥18 years on stable AHA step 1 diet.
3. For primary prevention, LDL > 130 mg/dL and for secondary prevention LDL>70 and <100mg/dL. .
4. CPK, ALT and AST < 1.5 x upper limit of normal at baseline.

Exclusion Criteria:

1. Women currently receiving cyclical hormones.
2. Treatment with hypolipidemic drugs during the last month.
3. Oral corticosteroids, NSAID, COX-1 inhibitors and other antiplatelet drugs.
4. Women with childbearing potential unless on safe contraception.
5. Psychiatric disease with defect in judgement.
6. Severe renal or hepatic diease.
7. Uncontrolled hypo- or hyperthyroidism.
8. Contraindication for ezetimibe or statin treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-07; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Spearsman's correlation coefficients will be calculated to determine the relation between changes in lipid parameters and changes in LDL tendency to oxidation and platelet aggregation.

CONTACTS AND LOCATIONS:
Overall Officials: Osamah Hussein, MD, Principal Investigator — Internal Medicine Department A, Ziv Medical Center
Locations (1):
- Internal Medicine Department A ,Ziv Goverment Hospital, Safed, Israel

REFERENCES:
- [Background] Sanderson S, Emery J, Baglin T, Kinmonth AL. Narrative review: aspirin resistance and its clinical implications. Ann Intern Med. 2005 Mar 1;142(5):370-80. doi: 10.7326/0003-4819-142-5-200503010-00012. PMID 15738456
- [Background] Kamath S, Blann AD, Lip GY. Platelet activation: assessment and quantification. Eur Heart J. 2001 Sep;22(17):1561-71. doi: 10.1053/euhj.2000.2515. No abstract available. PMID 11492985
- [Background] Bruno A, McConnell JP, Mansbach HH 3rd, Cohen SN, Tietjen GE, Bang NU. Aspirin and urinary 11-dehydrothromboxane B(2) in African American stroke patients. Stroke. 2002 Jan;33(1):57-60. doi: 10.1161/hs0102.102010. PMID 11779889
- [Background] Mammen EF, Comp PC, Gosselin R, Greenberg C, Hoots WK, Kessler CM, Larkin EC, Liles D, Nugent DJ. PFA-100 system: a new method for assessment of platelet dysfunction. Semin Thromb Hemost. 1998;24(2):195-202. doi: 10.1055/s-2007-995840. PMID 9579642
- [Background] Jefferson BK, Foster JH, McCarthy JJ, Ginsburg G, Parker A, Kottke-Marchant K, Topol EJ. Aspirin resistance and a single gene. Am J Cardiol. 2005 Mar 15;95(6):805-8. doi: 10.1016/j.amjcard.2004.11.045. PMID 15757620
- [Background] Reilly MP, Pratico D, Delanty N, DiMinno G, Tremoli E, Rader D, Kapoor S, Rokach J, Lawson J, FitzGerald GA. Increased formation of distinct F2 isoprostanes in hypercholesterolemia. Circulation. 1998 Dec 22-29;98(25):2822-8. doi: 10.1161/01.cir.98.25.2822. PMID 9860782
- [Background] Patrono C. Aspirin resistance: definition, mechanisms and clinical read-outs. J Thromb Haemost. 2003 Aug;1(8):1710-3. doi: 10.1046/j.1538-7836.2003.00284.x. No abstract available. PMID 12911581
- [Background] Cipollone F, Ciabattoni G, Patrignani P, Pasquale M, Di Gregorio D, Bucciarelli T, Davi G, Cuccurullo F, Patrono C. Oxidant stress and aspirin-insensitive thromboxane biosynthesis in severe unstable angina. Circulation. 2000 Aug 29;102(9):1007-13. doi: 10.1161/01.cir.102.9.1007. PMID 10961965
- [Background] Surya II, Akkerman JW. The influence of lipoproteins on blood platelets. Am Heart J. 1993 Jan;125(1):272-5. doi: 10.1016/0002-8703(93)90096-r. No abstract available. PMID 8380241
- [Background] Ardlie NG, Selley ML, Simons LA. Platelet activation by oxidatively modified low density lipoproteins. Atherosclerosis. 1989 Apr;76(2-3):117-24. doi: 10.1016/0021-9150(89)90094-4. PMID 2730708
- [Background] Osamah H, Mira R, Sorina S, Shlomo K, Michael A. Reduced platelet aggregation after fluvastatin therapy is associated with altered platelet lipid composition and drug binding to the platelets. Br J Clin Pharmacol. 1997 Jul;44(1):77-83. doi: 10.1046/j.1365-2125.1997.00625.x. PMID 9241100
- [Background] CHIAMORI N, HENRY RJ. Study of the ferric chloride method for determination of total cholesterol and cholesterol esters. Am J Clin Pathol. 1959 Apr;31(4):305-9. doi: 10.1093/ajcp/31.4.305. No abstract available. PMID 13637038
- [Background] LOWRY OH, ROSEBROUGH NJ, FARR AL, RANDALL RJ. Protein measurement with the Folin phenol reagent. J Biol Chem. 1951 Nov;193(1):265-75. No abstract available. PMID 14907713